CLINICAL TRIAL: NCT06009783
Title: Real World Utility of ChatGPT in Pre-vasectomy Counselling in an Office-based Setting
Brief Title: Utility of ChatGPT in Pre-vasectomy Counselling in an Office-based Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, PremalPatel, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS25978 (H2023:136)
Record Dates: First submitted 2023-06-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Vasectomy; Contraception
Keywords: vasectomy; ChatGPT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm - ChatGPT (Experimental): Patient's interested in participating in the intervention group will be provided a secure ChatGPT account. They will have the opportunity to converse with ChatGPT to ask any potential questions they may have regarding their upcoming vasectomy. Patient's will then be seen for the standard pre-vasectomy consultation.
  Interventions: Other: ChatGPT Language Model
- Control arm - no ChatGPT (No Intervention): No intervention - standard of care

INTERVENTIONS:
Other: ChatGPT Language Model — ChatGPT Language Model - ability to converse with the model and ask questions regarding vasectomies
  Arms: Intervention arm - ChatGPT

SUMMARY:
The investigators wish to perform a pilot study at the Manitoba Men's Health Clinic to assess if pre-vasectomy counseling with ChatGPT can safely streamline the consultation process by reducing visit times, while increasing patient satisfaction with the consultation process.

DETAILED DESCRIPTION:
The release of ChatGPT, a natural language AI chat bot, has recently captured the attention of the general public and medical professionals world-wide. ChatGPT is a conversational AI language model designed by OpenAI that utilizes deep learning techniques to generate human like responses to questions. There has been increasing interest among the medical community on developing new ways to harness this technology to aid medical professionals. New applications have included writing scientific manuscripts, drafting correspondents, as well as testing its ability on standardized medical licensing examinations. ChatGPT was able to perform at or near passing threshold on the United States Medical Licensing Exam (USMLE). Despite ChatGPT demonstrating good medical knowledge, it is still unclear if this translates to real world clinical practice.

Physician burnout is becoming an increasing problem. Per a recent Canadian Urologic Association (CUA) census, burnout was identified in 39% of urologists, with high number of patient visits/week to be cited as a predictor predictive of burnout. That begs the question, can ChatGPT be used for patient counseling and to improve patient flow in one's practice? ChatGPT has been shown to provide effective and safe responses to medical questions and even "curbside" consultations. However its ability to counsel patients in real time has not yet been studied.

As such, the investigators wish to perform a pilot study at the Manitoba Men's Health Clinic to assess if pre-vasectomy counseling with ChatGPT can safely streamline the consultation process by reducing visit times, while increasing patient satisfaction with the consultation process. If the hypothesis provides true, further implementation of ChatGPT in a healthcare practice may work to reduce the burden on health care providers.

There are no predicted adverse events of this study. There are no identified potential harms of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vasectomies interested in participating
* Adult (>18 years old)
* Consenting

Exclusion Criteria:

* Do not consent, uninterested in participating

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Length of Consultation | Through study completion, estimated to be 2 months measured for each phone call
  Length of pre-vasectomy consultation as measured from beginning to end of telephone call
Number of questions asked | Through study completion, estimated to be 2 months measured for each phone call
  Number of questions asked during pre-vasectomy consultation
Satisfaction of patients assessed by Likert scale | Through study completion, estimated to be 2 months measured for each patient
  Satisfaction of patients as measured by questionnaire with 10-point Likert Scale ([0-10] higher score correlates with higher satisfaction)

SECONDARY OUTCOMES:
Commonly asked questions | Through study completion period, estimated to be 2 months
  Chat logs will be reviewed to examine common themes or questions and reported using descriptive statistics.
Incidence of inaccurate ChatGPT responses | Through study completion period, estimated to be 2 months
  ChatGPT responses will be reviewed by two licensed clinicians experienced in vasectomies to determine rates of inaccurate responses by the language models responses to patient questions. Incidence of inaccurate ChatGPT responses will be reported and through descriptive analysis this will be described and inaccurate responses will be conveyed.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Patel, MD, Principal Investigator — Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No